CLINICAL TRIAL: NCT03661099
Title: INtegrated Colonoscopy Improvement Program in Italy (INCIPIT)
Brief Title: INtegrated Colonoscopy Improvement Program in Italy
Acronym: incipit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Pier Alberto Testoni, MD, IRCCS San Raffaele
Other Study IDs: INCIPIT/2017
Record Dates: First submitted 2018-08-29; First posted 2018-09-07 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Colon Lesion; Colon Polyp
MeSH Terms: conditions — Colonic Polyps | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: colonoscopy — endoscopists' performance outcome

SUMMARY:
The Italian Society of Digestive Endoscopy (SIED) and the Italian Association of Gastroenterologists and Hospital Digestive Endoscopists (AIGO) want to develop an effective training program for endoscopists to improve the quality of colonoscopies through careful evaluation of quality indicators and how they can be improved with an appropriate educational program. Primary objective of this study is to evaluate the variation of "Polyp Detection Rate (PDR) and Adenoma Detection Rate (ADR)" obtained by operators at high and low volume of colonoscopy before and after a training period. Secondary objectives are to compare high and low volume endoscopists' performance before and after training comparing by evaluation of withdrawal time; Number polyps / patient and Number adenomas / patient; the percentage and time of intubation of the cecum, ; patient's pain perception based on the Nurse Assessed Patient Comfort Score (NAPCOMS) scale. The study is structured as follow:

* A first phase when all endoscopists collect the results of 200 colonoscopies in an electronic Case Report Form (eCRF) is formed(maximum enrollment period 4 months).
* A second phase of training through an e-platform in which the endoscopists are offered with an online refresh reviewing the international standard parameters to perform a quality colonoscopy. Once the final training exam have been passed, the endoscopist will be able to access the third phase
* A third phase in which the endoscopists will collect prospectively the colonoscopies they perform in an eCRF (maximum enrollment period 4 months).

ELIGIBILITY:
Inclusion Criteria:

* patients between 50 and 75 years old
* colonoscopy for cancer screening program, post polypectomy follow up, patients with abdominal symptoms suggestive for colonic pathology.

Exclusion Criteria:

* patients aged < 50 or > 75 yrs

  * presence of alarm symptoms
  * American Society of Anesthesiologists (ASA) Classification ≥ 3
  * presence of colonic stenosis
  * previous colonic resection
  * Presence of diverticulitis
  * history of Inflammatory Bowel Disease (IBD)
  * History of polyposis syndrome
  * Pregnancy or breastfeeding
  * inability to provide informed consent
  * Severe cardiovascular illness
  * contraindication to undergo to sedation
  * Anticoagulant therapy
  * Melanosis coli

Ages: 50 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient aged between 50 and 75 years old who present with abdominal symptoms suggestive for colonic patholgy or included in cancer screening program
Sampling Method: Non-Probability Sample
Enrollment: 21250 (Estimated)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 9 months
  to evaluate Adenoma Detection Rate obtained by operators at high and low volume of colonoscopy before and after a training period(ADR)"
Polyps detection rate | 9 months
  to evaluate the variation of "Polyp Detection Rate (PDR) obtained by operators at high and low volume of colonoscopy before and after a training period

SECONDARY OUTCOMES:
Withdrawal time | 9 months
  to evaluate the amount of time spent viewing during the withdrawal of the scope
Number polyps / patient | 9 months
  Number of polyps found in each patient
Number adenomas / patient | 9 months
  Number of adenomas found in each patient
percentage of intubation of the cecum | 9 months
  percentage of colonoscopy in which endoscopist reach cecum
time of intubation of the cecum | 9 months
  the amount of time spent by endoscopist to reach cecum
patient's pain perception assessed by Nurse Assessed Patient Comfort Score (NAPCOMS) | 9 months
  evaluate tolerability of colonoscopy. NAPCOMS includes 3 domains: pain, sedation, and a global subjective assessment of tolerability. The pain domain is defined by using the dimensions of intensity (0. None or minimal; 1 mild; 2. Moderate; 3 severe), frequency (0. None; 1. Few 1 or 2 episodes; 2. Several times (3-4 episodes); 3. Frequent); and duration (0. None; 1 short duration; 2 Moderate duration; 3 Long duration).
  Sedation is rated according to level of consciousness ranging from 0 (wide awake) to 3 (unconscious), whereas the global tolerability score is rated from 0 (very well tolerated) to 3 (poorly tolerated). The overall NAPCOMS was defined as the sum of the severity, frequency, and duration of pain domains. Level of sedation and overall global tolerability ratings were assessed separately A NAPCOMS of 6 or greater corresponded with a patient rating of moderate to severe discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Pier Alberto Testoni, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided